CLINICAL TRIAL: NCT06650631
Title: The Effectiveness of Heat Treatment on Knee Pain in Patients With Osteoarthritis - an International, Multicenter Clinical Investigation. Prospective, Open-label, One-arm, Post-market, Effectiveness Clinical Investigation
Brief Title: The Effectiveness of Heat Treatment on Knee Pain in Patients With Osteoarthritis - an International, Multicenter Clinical Investigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161(B)MD22324
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-10

CONDITIONS: Pain Management; Osteoarthritis
Keywords: Pain; Osteoarthritis; ThermaCare®; Medical Device
MeSH Terms: conditions — Agnosia; Osteoarthritis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group: Patients with moderate knee osteoarthritis (Experimental): Patient without acute flares or inflammation enrolled. The overall duration of the investigation is expected to be 11 days, including screening days. The maximum treatment duration for each patient is 7 days (8h/d)
  Interventions: Device: Knee Heatwraps

INTERVENTIONS:
Device: Knee Heatwraps — To treat the painful knee joint in patients with osteoarthritis without acute flares or inflammation. The investigational device will be used in accordance with the Instructions for Use.

SUMMARY:
This post-market clinical follow-up, open-label, multicenter clinical investigation is designed to investigate the effectiveness, safety and tolerability of ThermaCare® Knee Heatwraps in the painful knee joint due to osteoarthritis. Approximately 80 patients, 19-69 years old inclusive, with moderate knee osteoarthritis (without acute flares or inflammation) will be enrolled. The overall duration of the investigation is expected to be 11 days, including screening days. The maximum treatment duration for each patient is 7 days (8h/d).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before inclusion in the investigation.
* Any gender, any ethnic origin, 19-69 years old inclusive.
* Body Mass Index 18.5-40 kg/m2 inclusive.
* Full comprehension: ability to comprehend the full nature and purpose of the clinical investigation.
* Patient with diagnosis of mono or bilateral moderate knee osteoarthritis with knee pain intensity > 40 mm on a 0-100 mm VAS, able to independently ambulate without walking aid.
* Availability of a radiography of the selected knee not older than 6 months.
* Patient is either not of childbearing potential or must agree not to start a pregnancy from the signature of the informed consent up to the final visit

Exclusion Criteria:

* Clinically significant abnormal physical findings which could interfere with the objectives of the investigation
* History of anaphylaxis to drugs or allergic reactions in general, which could affect the outcome of the clinical investigation.
* Significant history of diseases that may interfere with the aim of the clinical investigation.
* History of (in the last 6 months) or ongoing intra-articular injection involving the selected knee. History of ongoing physical therapy involving the selected knee.
* Presence of flares, inflammation, effusion and swelling at the selected knee.
* Any skin injury, wound, irritation, rash, bump, sore and/or discoloration at the application area.
* Surgery at the selected knee in the 12 months preceding the clinical investigation.
* Any medication that could interfere with the investigation procedures or investigation outcome.
* Use of other hot or cold therapies for the selected knee.
* Positive pregnancy test at screening; pregnant or breastfeeding women
* History of (within the past 12 months) or current drugs or alcohol abuse
* Individuals unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced because of a compromised position, expectation of benefits or fear of retaliatory response.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At home from Day 1 to Day 4.
  The primary endpoint of this clinical investigation is the change from baseline of pain intensity measured by Visual Analogue Scale (VAS) at Day 4, i.e., after 3 days of treatment.
  The VAS was chosen for the pain evaluation since it is a simple, quick and easy to use scale, suitable for different populations, such as adults and elderly individuals.
  Pain intensity will be measured using a 0-100 mm VAS.

SECONDARY OUTCOMES:
Sensorial perceptions evaluation | At 15, 30, 45 min, 1 and 4 h post-application on Day 1
  Results of the sensorial perceptions evaluation collected by a questionnaire. Questionnaire replies will be self-recorded by the patients in their individual diaries.
Pain intensity measured (%) | At 8 and 16 h post-application; From Day 1 to Day 7
  Percent change and change from baseline of pain intensity measured by VAS. The Visual Analogue Scale was chosen for the pain evaluation since it is a simple, quick and easy to use scale, suitable for different populations, such as adults and elderly individuals.
Functional levels and joint health measured (%) | At 8 day (final visit)
  Percent change and change from baseline in functional levels and joint health measured by Knee Injury and Osteoarthritis Outcome (KOOS) questionnaire at final visit.
  The questionnaire is an established patient-reported outcome instrument commonly used in clinical research. It is utilized to measure the changes in patient's health status in a standardized way. The questionnaire was chosen since adequate to both older and younger patients, able to combine short and long-term outcomes in a meaningful way and self-administered to patients through a questionnaire. The format is user-friendly and it takes about 10 minutes to fill-in. The standard KOOS questionnaire foresees 5 dimensions: pain, symptoms, activity of daily living, sport and recreation, quality of life. The sport, recreation dimension will not be assessed in this clinical investigation because we expect the enrolment of many elderly patients, for whom this section would not be applicable. The pain is already evaluatedby VAS.
Health status evaluation | At final visit (Day 8).
  Results of the overall health status evaluation performed by the Investigator by the CGI-I scale (Clinical Globally Impression - Improvement).
  This scale was selected since it is a simple, brief and stand-alone method allowing the clinician to assessing treatment response and overall improvement or worsening of the health conditions in clinical study participants.
  Sensorial perceptions and subject's satisfaction will be evaluated using questionnaires specifically designed for this purpose for this clinical investigation.
  CGI-I scale including 7 levels of achieved improvement/worsening (final visit/ETV).
Safety evaluation | From day 0 to day 8.
  Adverse events (AEs), including serious adverse events/serious device effects and special situations.
  Device deficiencies that might have led to a serious adverse event and any new findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Ars Medica Clinic, Gravesano, Switzerland, Switzerland